CLINICAL TRIAL: NCT01506908
Title: Evaluation of the Nicotine Mini Lozenge in Relief of Provoked Acute Craving
Brief Title: Provoked Craving Assessment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S7121359
Record Dates: First submitted 2011-12-15; First posted 2012-01-10 (Estimated); Results first posted 2014-01-30 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Smoking Dependence; Smoking
Keywords: craving
MeSH Terms: conditions — Smoking | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine Polacrilex mint mini lozenge (Active Comparator)
  Interventions: Drug: oral nicotine
- placebo (Placebo Comparator): mint mini lozenge with no active
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: oral nicotine — oral nicotine replacement product
  Arms: Nicotine Polacrilex mint mini lozenge
Drug: Placebo — no active
  Arms: placebo

SUMMARY:
Evaluation of the ability of a nicotine mini lozenge to provide early relief of craving for a cigarette in smokers

ELIGIBILITY:
Inclusion Criteria:

* Current cigarette smokers who have smoked regularly, and smoke more than 20 cigarettes per day on a regular basis for at least a year;
* Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history.

Exclusion Criteria:

* Any disease that may interfere with the absorption, metabolism or excretion of the study product.
* A medical condition that might jeopardise the safety of the subject or the validity of the study results. For example, recent myocardial infarction or cerebrovascular incident (within 12 weeks of the screening visit), phenylketonuria, unstable or worsening angina pectoris, Prinzmetals angina or severe cardiac arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Los Angeles Clinical Trials, Burbank, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=19927

REFERENCES:
- [Derived] Nides M, Shanga GM, Bishop A, Becker WD. Nicotine Lozenges in the Relief of Behaviorally Provoked Craving. Am J Health Behav. 2018 May 1;42(3):69-80. doi: 10.5993/AJHB.42.3.7. PMID 29663982

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Of 423 screened participants, 323 were randomized while 94 did not meet the study criterion and remaining 6 discontinued due to other reasons. All randomized participants had a history of smoking more than 20 cigarettes per day.
Groups:
- Nicotine Lozenge 4 Milligrams (mg): Participants received a single dose of 4 mg nicotine polacrilex mint lozenge, through oral route.
- Matched Placebo: Participants received a single dose of matched placebo mint lozenge, through oral route.
Period: Overall Study
Arm/Group | Nicotine Lozenge 4 Milligrams (mg) | Matched Placebo
Started | 162 | 161
Completed | 161 | 161
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nicotine Lozenge 4 mg: Participants received a single dose of 4 mg nicotine polacrilex mint lozenge, through oral route.
- Total: Total of all reporting groups
Arm/Group | Nicotine Lozenge 4 mg | Matched Placebo | Total
Number analyzed (Participants) | 162 | 161 | 323
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.69 (12.13) | 44.45 (11.64) | 44.07 (11.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 74 | 149
  Male | 87 | 87 | 174
Body Mass Index [Mean (Standard Deviation); unit: Kilograms (kg)/ meter (m)^2] | 27.79 (3.73) | 27.56 (4.05) | 27.67 (3.89)

OUTCOME MEASURES:

1. Primary Outcome: Change From Post-cue Baseline in Nicotine Craving Score at 5 Minutes
Description: Participants completed a nicotine craving assessment consisting of following five items: I have a desire for a cigarette right now, if it were possible I would smoke right now, All I want right now is a cigarette, I have an urge for a cigarette, I crave a cigarette right now. All participants indicated their craving intensity on a pre-drawn 100 mm scale ranging from 0 (disagree) to 100 (agree). At the end of the craving assessment period, mean VAS score was measured.
Time Frame: Post-cue baseline,5 minutes
Population: Intention to Treat (ITT) population: All randomized participants who had at least one cravings assessment measurement post dose. The imputation of missing craving score was based on last observation carried forward (LOCF) technique.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Nicotine Lozenge 4 mg | Matched Placebo
Number analyzed (Participants) | 162 | 161
Score on a scale | -41.8 [-45.8 to -37.7] | -25.9 [-30.0 to -21.8]
Statistical Analysis 1: Comparison: Nicotine Lozenge 4 mg vs Matched Placebo; Null hypothesis considered the population's change from post-cue baseline in craving score mean to be equal in both treatment groups at 5 minutes; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least squares means difference = -15.9, 95% CI 2-sided [-21.6 to -10.2] — Treatment comparisons were made between 4 mg nicotine lozenge and placebo lozenge at 5% significance level

2. Secondary Outcome: Change From Post-cue Baseline in Nicotine Craving Score at 1 Minute
Description: as for outcome 1
Time Frame: Post-cue baseline, 1 minute post treatment administration
Population: ITT population: All randomized participants who had at least one cravings assessment measurement post dose. The imputation of missing craving score was based on LOCF technique.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Nicotine Lozenge 4 mg | Matched Placebo
Number analyzed (Participants) | 162 | 161
Score on a scale | -17.2 [-20.1 to -14.2] | -12.9 [-15.9 to -10.0]
Statistical Analysis 1: Comparison: Nicotine Lozenge 4 mg vs Matched Placebo; Null hypothesis considered the population's change from post-cue baseline in craving score mean to be equal in both treatment groups at 1 minute; Test type: Superiority or Other; p = 0.0511, ANCOVA; Least squares means difference = -4.2, 95% CI 2-sided [-8.4 to 0.0] — Treatment comparisons were made between 4 mg nicotine lozenge and placebo lozenge at 5% significance level

3. Secondary Outcome: Change From Post-cue Baseline in Nicotine Craving Score at 3 Minutes
Description: as for outcome 1
Time Frame: Post-cue Baseline, 3 minutes post treatment administration
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Nicotine Lozenge 4 mg | Matched Placebo
Number analyzed (Participants) | 162 | 161
Score on a scale | -31.1 [-34.8 to -27.5] | -19.6 [-23.2 to -15.9]
Statistical Analysis 1: Comparison: Nicotine Lozenge 4 mg vs Matched Placebo; Null hypothesis considered the population's change from post-cue baseline in craving score mean to be equal in both treatment groups at 3 minutes; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least squares means difference = -11.6, 95% CI 2-sided [-16.7 to -6.4] — Treatment comparisons were made between 4 mg nicotine lozenge and placebo lozenge at 5% significance level

4. Secondary Outcome: Change From Post-cue Baseline in Nicotine Craving Score at 7 Minutes
Description: as for outcome 1
Time Frame: Post-Cue Baseline, 7 minutes post treatment administration
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Nicotine Lozenge 4 mg | Matched Placebo
Number analyzed (Participants) | 162 | 161
Score on a scale | -48.2 [-52.5 to -43.9] | -30.5 [-34.8 to -26.2]
Statistical Analysis 1: Comparison: Nicotine Lozenge 4 mg vs Matched Placebo; Null hypothesis considered the population's change from post-cue baseline in craving score mean to be equal in both treatment groups at 7 minutes; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least squares means difference = -17.8, 95% CI 2-sided [-23.8 to -11.7] — Treatment comparisons were made between 4 mg nicotine lozenge and placebo lozenge at 5% significance level

5. Secondary Outcome: Change From Post-cue Baseline in Nicotine Craving Score at 10 Minutes
Description: as for outcome 1
Time Frame: Post-Cue Baseline, 10 minutes post treatment administration
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Nicotine Lozenge 4 mg | Matched Placebo
Number analyzed (Participants) | 162 | 161
Score on a scale | -50.8 [-55.3 to -46.2] | -32.9 [-37.5 to -28.3]
Statistical Analysis 1: Comparison: Nicotine Lozenge 4 mg vs Matched Placebo; Null hypothesis considered the population's change from post-cue baseline in craving score mean to be equal in both treatment groups at 10 minutes; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least square mean difference = -17.9, 95% CI 2-sided [-24.4 to -11.4] — Treatment comparisons were made between 4 mg nicotine lozenge and placebo lozenge at 5% significance level

6. Secondary Outcome: Number of Participants With Adverse Events (AEs), Treatment Related AEs, and Serious AEs (SAEs)
Description: AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with study treatment/s. Treatment related AE was defined as any AE considered to be possibly, probably or highly probably related to study medication. SAE was defined as any untoward medical occurrence that at any dose results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization results in disability/ incapacity; is a congenital anomaly/ birth defect.
Time Frame: Baseline to Day 5 post treatment administration
Population: Safety population: All randomized participants who received the study treatments were considered evaluable for safety.
Measure: Number; unit: Participants
Arm/Group | Matched Placebo | Nicotine Lozenge 4 mg
Number analyzed (Participants) | 161 | 162
Participants
  AEs | 12 | 54
  Treatment Related AEs | 11 | 54
  SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events encountered or spontaneously reported following administration of any investigational product (including washout product), or for up to 5 days after the last administration of investigational product were recorded.
Groups:
- Placebo Lozenge: Participants received a single dose of matched placebo mint lozenge, through oral route.
Arm/Group | Nicotine Lozenge 4 mg | Placebo Lozenge
Serious Adverse Events (participants affected / at risk) | 0/162 | 0/161
Other Adverse Events (participants affected / at risk) | 54/162 | 12/161
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Lozenge 4 mg (N=162) | Placebo Lozenge (N=161)
Nausea (Gastrointestinal disorders) | 24 (24) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 3 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Heart Rate Increased (Investigations) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.